CLINICAL TRIAL: NCT04888546
Title: A Single-arm, Multicenter Phase Ib Clinical Trial of the Efficacy and Safety of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule Neoadjuvant in the Treatment of Resectable Hepatocellular Carcinoma With a High Risk of Recurrence or Metastasis
Brief Title: TQB2450 Combined With Anlotinib Hydrochloride in the Perioperative Treatment of Hepatocellular Carcinoma Hydrochloride Neoadjuvant Therapy for Resectable Hepatocellular Carcinoma With a High Risk of Recurrence or Metastasis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hong Zhao, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-Ib-13
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Patients With Resectable Hepatocellular Carcinoma Who Are at High Risk of Recurrence or Metastasi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib hydrochloride capsules combined with TQB2450 injection (Other): Anlotinib hydrochloride capsules (10mg po qd, Two weeks off for one week) combined with TQB2450 injection (1200mg ivgtt, q3W)
  Interventions: Drug: Anlotinib hydrochloride capsules＋ TQB2450 injection

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsules＋ TQB2450 injection — Anlotinib hydrochloride capsules is a new type of small molecule multi-target tyrosine kinase inhibitor against angiogenesis.
  TQB2450 is a humanized monoclonal antibody targeting PD-L1, which prevents PD-L1 from binding to the PD-1 and B7.1 receptors on the surface of T cells, so as to restore the activity of T cells and thereby enhance the immune response, and has the potential to treat various types of tumors.

SUMMARY:
In this study, single cell transcriptome sequencing will be performed on the tissue samples punctured and the surgically resected specimens to explore the gene mutation sites related to efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent;
2. Age: 18-75 years old;ECOG PS：0-1；The expected survival is more than 6 months;
3. No gender limitation;
4. Histologically confirmed hepatocellular carcinoma;
5. Meet resectable surgical criteria;
6. Child-Pugh:A or B;
7. According to RECIST 1.1, there is at least one evaluable lesion that has not been treated;

Exclusion Criteria:

1. Fibrolamellar HCC, sarcomatoid HCC, or mixed bile duct cell-HCC is known to exis;
2. Preoperative systemic treatment including chemotherapy, targeted therapy and immunotherapy;Preoperative local treatment including radiotherapy, interventional therapy and ablative therapy;
3. No radical resection could be performed after adequate imaging evaluation;
4. Present or present with other malignant tumors within 3 years.Two conditions were eligible for inclusion: 5 consecutive years of disease-free survival (DFS) for other malignancies treated with a single operation;Cured carcinoma in situ of the cervix, non-melanoma skin cancer, and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basement membrane)]; 5 . There are many factors that affect oral medications (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);

6. Hepatitis B combined with hepatitis C; 7. Patients with portal hypertension have high bleeding risk considered by the researcher, or gastroscopy or gastroscopy confirmed red signs, or gastroscopy found active ulcers with high bleeding risk;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | 6 months
  No histologic evidence of malignancy or only the ingredients of carcinoma in situ was found in primary tumors.
Overall response rate (ORR) | through study completion, an average of 6 months
  Objective response rate refers to the percentage of complete (CR) or partial response (PR) subjects determined by the investigator based on RECIST 1.1 .

SECONDARY OUTCOMES:
Progression free survival(PFS) | through study completion, an average of 1 year
  Disease control rate refers to the percentage of subjects with a disease stabilization (SD) of 6 weeks or greater in complete response, partial response, or at least 6 weeks, as determined by RECIST 1.1.
Overall survival (OS) | through study completion, an average of 1 year
  It is defined as the time from randomization to death from any cause during the course of the study
The incidence and severity of AE | through study completion, an average of 1 year
  AE is any adverse medical event that occurs in a subject participating in a clinical trial that may or may not have a causal relationship with the treatment.An AE can be any adverse and unexpected signs (including abnormal laboratory results), symptoms, or diseases that are time-related to the use of the study drug, whether or not the study drug is considered relevant.
The incidence and severity of SAE | through study completion, an average of 1 year
  When subjects were tested with drug adverse events of comply with the following one or more than a standard as a serious adverse event (SAE) : death, life-threatening, permanent or severe disability or loss of function, subjects requiring hospitalization or extend the length of hospital stay, congenital anomaly, or birth defects, subsequent pregnancy happen (natural or artificial abortion, the pregnancy is terminated because of medical reasons) and other important medical event (no threat to life or death, but may endanger patients or may lead to interventions are needed to prevent this happen).

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China